CLINICAL TRIAL: NCT04582721
Title: PREFerred Neurostimulation MODdalities to Treat Chronic Intractable Back Pain, A 3x3 Crossover Study
Brief Title: PREFerred Neurostimulation MODdalities - PREFMOD Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale Regionale di Lugano (Other)
Collaborators: Paolo Maino MD PhD, Sponsor Investigator (Unknown)
Responsible Party: Principal Investigator, Eva Koetsier MD PhD LLM, MD PhD LLM, Ospedale Regionale di Lugano
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NSI-TD-010
Record Dates: First submitted 2019-07-25; First posted 2020-10-09 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CON-SCS with subcutaneous stimulation (Active Comparator): 7 days Conventional Spinal Cord Stimulation with subcutaneous stimulation
  Interventions: Other: Implantable Neurostimulator System (Spectra WaveWriter™ Spinal Cord Stimulator System), (Boston Scientific Neuromodulation Corporation, Valencia, California (CA), USA)
- HF-SCS (Active Comparator): 7 days High Frequency Spinal Cord Stimulation
  Interventions: Other: Implantable Neurostimulator System (Spectra WaveWriter™ Spinal Cord Stimulator System), (Boston Scientific Neuromodulation Corporation, Valencia, California (CA), USA)
- Combination Therapy (Active Comparator): 7 days a combination of CON-SCS with subcutaneous stimulation and HF-SCS
  Interventions: Other: Implantable Neurostimulator System (Spectra WaveWriter™ Spinal Cord Stimulator System), (Boston Scientific Neuromodulation Corporation, Valencia, California (CA), USA)

INTERVENTIONS:
Other: Implantable Neurostimulator System (Spectra WaveWriter™ Spinal Cord Stimulator System), (Boston Scientific Neuromodulation Corporation, Valencia, California (CA), USA) — the participants with chronic intractable back or back and leg pain will be implanted with the stimulation lead(s). The leads are initially connected to an external trial neurostimulator. Patients will be implanted with two epidural leads and two subcutaneous leads. A three weeks trial phase will follow. The first two days after the leads implant will be without stimulation and thereafter alternating stimulation every week will start, randomly ordering the treatments using a Williams design balanced for first-order carryover effects (i.e. incorporating 6 different treatment orders), from:
  * 1) CON-SCS with Subcutaneous stimulation
  * 2) HF-SCS
  * 3) Combination Therapy A patient's favored SCS mode, providing that there is at least 50% reduction in pain intensity on the NRS in the trial phase, will then be implanted and patients will be followed up for 12 months.

SUMMARY:
This is a prospective 3x3 crossover study with randomized treatment order, comparing the short-term efficacy of conventional-spinal cord stimulation (CON-SCS) with subcutaneous stimulatio, high frequency-spinal cord stimulation (HF-SCS), and Combination Therapy, in patients with chronic intractable back pain (with or without leg pain).

DETAILED DESCRIPTION:
Patients will be preselected for inclusion in this study at the pain management center of Neurocenter of Southern Switzerland, Ente Ospedaliero Cantonale (EOC) Lugano, and will be informed about study-details by a study clinician. After informed consent signature, the participants with chronic intractable back or back and leg pain will be implanted with the stimulation lead(s). The leads are initially connected to an external trial neurostimulator. Patients will be implanted with two epidural leads and two subcutaneous leads. A three weeks trial phase will follow. The first two days after the leads implant will be without stimulation and thereafter alternating stimulation every week will start, randomly ordering the treatments using a Williams design balanced for first-order carryover effects (i.e. incorporating 6 different treatment orders), from:

* 1) CON-SCS with Subcutaneous stimulation
* 2) HF-SCS
* 3) Combination Therapy A patient's favored SCS mode, providing that there is at least 50% reduction in pain intensity on the NRS in the trial phase, will then be implanted and patients will be followed up for 12 months.

Pain intensity and pain medication will be assessed with a pain diary at baseline and during the trial phase and will be furthermore measured after 3, 6, and 12 months after the implantation. Physical functioning, Pain Extent, Patient Global Impression of Change (PGIC), and Satisfaction with stimulation treatment (SST) will be assessed during the trial phase and will be furthermore measured after 3, 6, and 12 months after the Implantable Nerve Stimulator (INS) implantation. The other secondary outcomes will be measured at baseline, and after 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at inclusion
* chronic, intractable back or back and leg pain during at least 6 months
* pain intensity of ≥ 5 on a NRS (ranging from 0 to 10)
* previous drug therapy unsuccessful

Exclusion Criteria:

* Psychological disorders
* Coagulation disorders
* Known immune-deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-04-09 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
back pain intensity | 21 days
  The difference in the intensity of back pain between the three neurostimulation modalities as measured by the numerical rating scale (NRS) from 0 to 10, where 0 is not pain and 10 is the maximum pain the person can experience, assessed at baseline and in the trial phase 21 days

CONTACTS AND LOCATIONS:
Locations (1):
- Centro del Dolore, Neurocentro, Opedale Regionale di Lugano, Lugano, Canton Ticino, Switzerland